CLINICAL TRIAL: NCT07122193
Title: A Phase 3, Randomized, Parallel-Group, Double-Blind, Multicenter Study Investigating the Safety and Efficacy of NT 201 Compared With Placebo in Adult Participants With Moderate to Severe Platysma Prominence in the United States
Brief Title: A Study of NT 201 in Adults With Moderate to Severe Platysma Prominence in the United States
Acronym: PLATINUM US
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NT-PPR-US001
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Neuromuscular Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Acetylcholine Release Inhibitors; Membrane Transport Modulators; Molecular Mechanisms of Pharmacological Action; Cholinergic Agents; Neurotransmitter Agents; incobotulinumtoxinA; Botulinum Toxins, Type A
Keywords: Platysma prominence
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Main Period: NT 201 (Experimental): Participants will receive NT 201 IM injection, once on Day 1 of the MP.
  Interventions: Drug: NT 201
- Main Period: NT 201 Matching Placebo (Placebo Comparator): Participants will receive NT 201 matching placebo IM injection, once on Day 1 of the MP.
  Interventions: Drug: NT 201 Placebo
- OLEX Period: NT 201 (Experimental): Participants will receive a reinjection of NT 201 IM injection, once on Day 1 of OLEX Cycle 1 and Cycle 2.
  Interventions: Drug: NT 201

INTERVENTIONS:
Drug: NT 201 — Clostridium Botulinum neurotoxin A (150 kiloDalton [kD], free of complexing proteins), powder for solution for injection.
  Other Names: IncobotulinumtoxinA; Xeomin/Bocouture; Xeomin Cosmetic; Xeomeen
  Arms: Main Period: NT 201; OLEX Period: NT 201
Drug: NT 201 Placebo — NT 201 matching-placebo
  Arms: Main Period: NT 201 Matching Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of NT 201 compared with placebo in participants with moderate to severe platysma prominence. The study will be conducted in two periods: Main Period (MP) and Open label Extension Period (OLEX).

ELIGIBILITY:
Inclusion Criteria:

* Presence of four (medial and lateral, left and right) platysmal bands assessed at screening and baseline.
* A score of Grade 3 ('moderate') or Grade 4 ('severe') on the MAPS-D at maximum contraction by the investigator and participant.

Exclusion Criteria:

* Hypersensitivity or a history of allergic reaction to botulinum toxin of any serotype or any of their formulation ingredients.
* Any medical condition that may put the participant at increased risk with exposure to botulinum toxin of any serotype, or any disorders that might interfere with neuromuscular function.
* Any serious disease or disorder that could interfere with the safe completion of treatment or with study outcome assessments, or compromise participant safety.
* Botulinum toxin treatment in the face (below the lower orbital rim), jawline, or neck within the last seven months.
* History of lower face surgery, neck or chest surgery, aesthetic procedures, and orthodontic procedures in the past 12 months.
* Planned surgery or aesthetic procedures to the lower face, neck, or chest during the study period.
* Anticipated need for treatment with botulinum toxin of any serotype for any indication during the study (other than study products).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Composite Achievement of Grade 1 or Grade 2 and at Least a 2-Grade Improvement From Baseline Based on Both the Investigator's Assessment and Participant's Self-Assessment Using the Merz Aesthetics Platysma Scale - Dynamic (MAPS-D) At Week 2 of MP | At Week 2 of MP
  MAPS-D is a validated five-point scale that will be used to grade the platysma prominence. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe). A lower score indicates improvement.

SECONDARY OUTCOMES:
Achievement of Grade 1 (None to Minimal) or Grade 2 (Mild) And at Least a 2-Grade Improvement From Baseline Based on the Investigator's Assessment Using MAPS-D at Week 2 of MP | At Week 2 of MP
  MAPS-D is a validated five-point scale that will be used to grade the platysma prominence. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe). A lower score indicates improvement.
Achievement of Grade 1 (None to Minimal) or Grade 2 (Mild) And at Least a 2-Grade Improvement From Baseline Based on the Participant's Self-Assessment Using MAPS-D at Week 2 of MP | At Week 2 of MP
  MAPS-D is a validated five-point scale that will be used to grade the platysma prominence. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe). A lower score indicates improvement.
Achievement of at Least a +1 (Somewhat Satisfied) Score Using the Participant's Satisfaction Questionnaire at Week 2 of MP | At Week 2 of MP
  Participants satisfaction questionnaire responses will be rated on a scale ranging from +3 (very satisfied) to -3 (very dissatisfied). A higher score indicates satisfaction.
Achievement of Grade 1 (None to Minimal) or Grade 2 (Mild) And at Least a 2-Grade Improvement From Baseline Based on Both the Investigator's Assessment and Participant's Self-Assessment Using MAPS-D at Week 1 and Week 4 up to Week 17 of MP | At Week 1 and Week 4 up to Week 17 of MP
  MAPS-D is a validated five-point scale that will be used to grade the platysma prominence. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe). A lower score indicates improvement.
Achievement of Grade 1 (None to Minimal) or Grade 2 (Mild) And at Least a 2-Grade Improvement From Baseline Based on the Investigator's Assessment Using MAPS-D at Week 1 and Week 4 up to Week 17 of MP | At Week 1 and Week 4 up to Week 17 of MP
  MAPS-D is a validated five-point scale that will be used to grade the platysma prominence. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe). A lower score indicates improvement.
Achievement of Grade 1 (None to Minimal) or Grade 2 (Mild) And at Least a 2-Grade Improvement From Baseline Based on Participant's Self-Assessment Using MAPS-D at Week 1 and Week 4 up to Week 17 of MP | At Week 1 and Week 4 up to Week 17 of MP
  MAPS-D is a validated five-point scale that will be used to grade the platysma prominence. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe). A lower score indicates improvement.
Achievement of at Least a +1 (Improved) Score on the Global Aesthetic Improvement Scale (GAIS)-Platysmal Bands Based on the Investigator's Assessment at Week 2 of MP | At Week 2 of MP
  GAIS is a balanced seven-point Likert scale (range -3 [very much worse] to +3 [very much improved]) commonly used in aesthetic medicine to rate post-treatment improvement in appearance. A higher score indicates improvement.
Achievement of at Least a +1 (Improved) Score on the GAIS-Platysmal Bands Based on the Participant's Self-Assessment at Week 2 of MP | At Week 2 of MP
  GAIS is a balanced seven-point Likert scale (range -3 [very much worse] to +3 [very much improved]) commonly used in aesthetic medicine to rate post-treatment improvement in appearance. A higher score indicates improvement.
Achievement of at Least a +1 (Improved) Score Using the GAIS-Lower Face Contour According to the Investigator's Assessment at Week 2 of MP | At Week 2 of MP
  GAIS is a balanced seven-point Likert scale (range -3 [very much worse] to +3 [very much improved]) commonly used in aesthetic medicine to rate post-treatment improvement in appearance. A higher score indicates improvement.
Achievement of at Least a +1 (Improved) Score Using the GAIS-Lower Face Contour According to the Participant's Self-Assessment at Week 2 of MP | At Week 2 of MP
  GAIS is a balanced seven-point Likert scale (range -3 [very much worse] to +3 [very much improved]) commonly used in aesthetic medicine to rate post-treatment improvement in appearance. A higher score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (26):
- United States (25):
  - Merz Investigative Site, Scottsdale, Arizona
  - Merz Investigative Site, Encino, California
  - Merz Investigative Site, Los Angeles, California
  - Merz Investigative Site, Redondo Beach, California
  - Merz Investigative Site, Santa Monica, California
  - Merz Investigative Site, Vista, California
  - Merz Investigative Site, Greenwood Village, Colorado
  - Merz Investigative Site, Westport, Connecticut
  - Merz Investigative Site, Washington D.C., District of Columbia
  - Merz Investigative Site, Aventura, Florida
  - Merz Investigative Site, Boca Raton, Florida
  - Merz Investigative Site, Bradenton, Florida
  - Merz Investigative Site, Coral Gables, Florida
  - Merz Investigative Site, West Palm Beach, Florida
  - Merz Investigative Site, Alpharetta, Georgia
  - Merz Investigative Site, Naperville, Illinois
  - Merz Investigative Site, Hunt Valley, Maryland
  - Merz Investigative Site, Mount Kisco, New York
  - Merz Investigative Site, New York, New York
  - Merz Investigative Site, Chapel Hill, North Carolina
  - Merz Investigative Site, Wilmington, North Carolina
  - Merz Investigative Site, Ardmore, Pennsylvania
  - Merz Investigative Site, Nashville, Tennessee
  - Merz Investigative Site, Dallas, Texas
  - Merz Investigative Site, Arlington, Virginia
- Merz Investigative Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No